CLINICAL TRIAL: NCT05135208
Title: Optimized Camera-based Patient Positioning in CT: Impact on Radiation Exposure.
Brief Title: Optimized Camera-based Patient Positioning in CT
Status: Completed | Type: Observational
Sponsor: Dr. Panagiota Manava (Other)
Responsible Party: Sponsor-Investigator, Dr. Panagiota Manava, Dr. med. Panagiota Manava, MD, Attending Radiologist, Principal Invesigator, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: CT_2021
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Radiation Dosage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: patients positioned with 3D camera
- control group: patients positioned by experienced radiology assistants

SUMMARY:
To evaluate the effect on radiation dose using intelligent camera positioning in comparison to manual positioning by the radiology assistant.

DETAILED DESCRIPTION:
The positioning of the patient at the beginning of every CT examination has an major influence on the image quality and especially on the respective effective patient dose in the CT scan. If the patient position is closer to the X-ray tube, the patient dose increases significantly and if the vertical patient position is chosen too far away from the X-ray tube, the applied dose decreases, but also the image quality.

In a retrospective observational study, patients were examined on the CT scanner Somatom X.Cite and divided into two groups, one group was with intelligent camera positioning and the other with manual positioning.

The patients received their CT scan at the Institute Radiology and Nuclear Medicine at the Nuremberg North Hospital strictly according to the clinical indication and without influence of the study.

ELIGIBILITY:
Inclusion Criteria:

Only patients with a clinical indication for a CT Scan

Exclusion Criteria:

renal insufficiency, manifest hyperthyroidism and pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 3118 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Effective dose | 10 months
  the absorbed dose to different organs of the body

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Lell, Prof. Dr., Study Director — Department of Radiology and Nuclear Medicine, Klinikum Nuernberg, Paracelsus Medical University, Germany
Locations (1):
- Institute of Radiology and Nuclear Medicine, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Booij R, Budde RPJ, Dijkshoorn ML, van Straten M. Accuracy of automated patient positioning in CT using a 3D camera for body contour detection. Eur Radiol. 2019 Apr;29(4):2079-2088. doi: 10.1007/s00330-018-5745-z. Epub 2018 Oct 10. PMID 30306328
- [Background] Kaasalainen T, Palmu K, Reijonen V, Kortesniemi M. Effect of patient centering on patient dose and image noise in chest CT. AJR Am J Roentgenol. 2014 Jul;203(1):123-30. doi: 10.2214/AJR.13.12028. PMID 24951205
- [Background] Saltybaeva N, Schmidt B, Wimmer A, Flohr T, Alkadhi H. Precise and Automatic Patient Positioning in Computed Tomography: Avatar Modeling of the Patient Surface Using a 3-Dimensional Camera. Invest Radiol. 2018 Nov;53(11):641-646. doi: 10.1097/RLI.0000000000000482. PMID 29762259
- [Background] Marsh RM, Silosky MS. The effects of patient positioning when interpreting CT dose metrics: A phantom study. Med Phys. 2017 Apr;44(4):1514-1524. doi: 10.1002/mp.12137. Epub 2017 Mar 17. PMID 28133763
- [Background] Dane B, O'Donnell T, Liu S, Vega E, Mohammed S, Singh V, Kapoor A, Megibow A. Radiation dose reduction, improved isocenter accuracy and CT scan time savings with automatic patient positioning by a 3D camera. Eur J Radiol. 2021 Mar;136:109537. doi: 10.1016/j.ejrad.2021.109537. Epub 2021 Jan 12. PMID 33454459
- [Derived] Manava P, Galster M, Ammon J, Singer J, Lell MM, Rieger V. Optimized Camera-Based Patient Positioning in CT: Impact on Radiation Exposure. Invest Radiol. 2023 Feb 1;58(2):126-130. doi: 10.1097/RLI.0000000000000904. Epub 2022 Aug 2. PMID 35926075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT05135208/Prot_SAP_000.pdf